CLINICAL TRIAL: NCT00122213
Title: An Individual-based Diet and Physical Activity Intervention Program to Prevent Accumulation of Abdominal Fat Mass in Recently Retired Men and Women
Brief Title: A Physical Activity and Diet Program to Prevent Accumulation of Abdominal Fat Mass in Recently Retired Men and Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Netherlands Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000T205
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Retirement; Weight Gain
Keywords: Prevention; Retirement; Physical activity; Diet; Weight gain; Body composition
MeSH Terms: conditions — Weight Gain; Motor Activity | interventions — Diet

INTERVENTIONS:
Behavioral: Behavior change on physical activity and diet

SUMMARY:
Advancing age in itself is associated with changes in body composition. However, during transitional life stages, such as retirement, detrimental changes on diet and physical activity may occur. This might lead to weight gain and accumulation of abdominal fat.

To prevent these changes, participants receive a low-intensity intervention on energy balance and related behaviours.

After six months, one and two years, the effects will be studied by comparing the intervention group with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy and recently retired

Exclusion Criteria:

* Using drugs that might influence body composition, digestion or physical activities

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Anthropometrics (body weight, height, circumferences, total body fat%, blood pressure)
Energy intake (Food Frequency Questionnaire)
Physical activity level (Physical Activity Scale for the Elderly)

SECONDARY OUTCOMES:
Psychosocial factors (attitude, social influence, self-efficacy etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Evert G Schouten, PhD, Study Chair — Wageningen University - Division of Human Nutrition

REFERENCES:
- [Derived] Werkman A, Hulshof PJ, Stafleu A, Kremers SP, Kok FJ, Schouten EG, Schuit AJ. Effect of an individually tailored one-year energy balance programme on body weight, body composition and lifestyle in recent retirees: a cluster randomised controlled trial. BMC Public Health. 2010 Mar 5;10:110. doi: 10.1186/1471-2458-10-110. PMID 20205704